CLINICAL TRIAL: NCT07304505
Title: An Open-Label Exploratory Analysis of Commercial Probiotics in Adults With Rheumatoid Arthritis
Brief Title: Probiotics in Adults With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ancilia Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AFCRO-201
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Microbiome; Probiotic
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): 6-week daily oral administration of Align Extra Strength Probiotic Supplement, produced by Procter & Gamble (Bifidobacterium longum subsp. longum 35624™)
  Interventions: Dietary Supplement: Align Extra Strength Probiotic Supplement

INTERVENTIONS:
Dietary Supplement: Align Extra Strength Probiotic Supplement — Bifidobacterium longum subsp. longum 35624™ (50mg): 5 x10^9 (5 billion) live bacteria per capsule

SUMMARY:
The goal of this clinical study is to collect data on the effect of probiotic administration on clinical outcomes in rheumatoid arthritis patients.

Participants will:

* Have a 6-week daily administration of a probiotic
* Collect fecal samples every other day during the first 3 weeks of the study and twice weekly over the last 3 weeks
* Visit the clinic at Baseline, Week 3 and Week 6 for checkup and testing

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be 18 years or older.
3. Clinical diagnosis of rheumatoid arthritis (RA) for more than 6 months.
4. Have been on stable RA treatment for 3 months and are expected to remain on stable RA treatment during the study.
5. Willing to consume the study product daily for the duration of the study.

Exclusion Criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
   2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that Participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.
   5. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
3. Has a history of drug and/or alcohol abuse.
4. Has food allergies or other issues with foods that would preclude intake of the Study Products including milk and soy allergies.
5. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results. Excluded health conditions include:

   1. history of mixed connective tissue disease or overlap syndrome (Systemic lupus erythematosus (SLE), Systemic sclerosis (scleroderma), Polymyositis/ dermatomyositis)
   2. Prior history or current inflammatory joint disease other than RA (such as psoriatic arthritis, gout, reactive arthritis, Lyme disease).
   3. Diagnosed gastrointestinal disease
   4. Gastrointestinal surgery, excluding cholecystectomy and appendectomy in the last five years.
   5. Renal failure
   6. Liver cirrhosis
6. Current or recent (in the past 8-weeks) use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

   a. Antibiotics
7. Current or recent (in the past 4-weeks) use of prohibited nutritional or non-nutritional supplements that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited supplements include:

   a. Probiotics
8. Current or recent (in the past 2-weeks) use of yoghurts containing probiotics.
9. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
10. Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Probiotic bacterial colonization | 6 weeks
  Change from baseline (Day 0) to Day 39 (including intermediate time points) in the relative abundance and/or detection frequency of the administered probiotic strain in stool

SECONDARY OUTCOMES:
RA clinical outcomes | 6 weeks
  Change from baseline (Day 0) to Day 21, and Day 39 on Rheumatoid Arthritis clinical outcomes as assessed by Clinical Disease Activity Index (CDAI) Total Score based on: Tender joint count, Swollen joint count, Patient Global disease Activity, Evaluator Global disease Activity. CDAI score is the sum of these components, ranging from 0 to 76, where higher scores are worse outcomes.

OTHER OUTCOMES:
Adverse events | 6 weeks
  Occurrence of any adverse events (AEs/SAEs) and/or changes in vital signs (Blood Pressure, Heart Rate, and Temperature) during probiotic administration

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No